CLINICAL TRIAL: NCT00538187
Title: Phase I Study of GX15-070 (NSC # 729280) and Bortezomib in Aggressive Relapsed/Recurrent Non-Hodgkin's Lymphoma
Brief Title: Obatoclax and Bortezomib in Treating Patients With Aggressive Relapsed or Recurrent Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00253; PHI-58; CDR0000566357; U01CA062505 (NIH)
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2013-05

CONDITIONS: Adult Non-Hodgkin Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obatoclax; Bortezomib

ARMS (1):
- Treatment (obatoclax mesylate, bortezomib) (Experimental): Patients will receive a 3-hour infusion of obatoclax and an infusion of bortezomib once a week for 4 weeks
  Interventions: Drug: obatoclax mesylate; Drug: bortezomib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: obatoclax mesylate — Given IV
  Other Names: GX15-070MS
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — correlative study
Other: pharmacological study — correlative study
  Other Names: pharmacological studies

SUMMARY:
Obatoclax may stop the growth of non-Hodgkin lymphoma by blocking blood flow to the cancer. Bortezomib and obatoclax may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving obatoclax together with bortezomib may kill more cancer cells. This phase I/II trial is studying the side effects and best dose of obatoclax when given together with bortezomib and to see how well they work in treating patients with aggressive relapsed or recurrent non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose of obatoclax mesylate when administered with bortezomib in patients with aggressive relapsed or recurrent non-Hodgkin lymphoma.

II. To describe the toxicities of this regimen at each dose studied in these patients.

III. To characterize the pharmacokinetic behavior of this regimen in these patients.

IV. To obtain preliminary information regarding the effect of obatoclax mesylate on several apoptotic regulatory pathways.

V. To document all clinical responses in these patients to this regimen.

OUTLINE: This is a multicenter study.

PHASE I: Patients receive obatoclax mesylate IV over 3 hours followed by bortezomib IV on days 1, 8, 15, and 22.

Treatment repeats every 35 days in the absence of disease progression or unacceptable toxicity. Pharmacokinetic evaluations of obatoclax mesylate are conducted in all patients during the first course.

PHASE II: Patients receive obatoclax mesylate IV over 3 hours followed by bortezomib IV on days 1, 8, 15, and 22 at the maximum tolerated dose determined in phase I.

Treatment repeats every 35 days for up to 1 year in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed relapsed or refractory non-Hodgkin lymphoma for which standard curative or palliative measures do not exist or are no longer effective, including any of the following subtypes:

  * Follicular grade I, II, or III lymphoma
  * Marginal zone lymphoma
  * Mantle cell lymphoma
  * Diffuse large B cell lymphoma
  * Small lymphocytic lymphoma
* Must have had at least one prior chemotherapeutic regimen:

  * Steroids or rituximab alone or local radiotherapy do not count as regimens
  * Tositumomab or ibritumomab tiuxetan allowed as regimens
* Clear evidence of disease progression or lack of response after the most recent therapy, including rituximab or local radiotherapy, is required
* At least 3 months since prior autologous stem cell transplantation and relapsed (>= 1 year since prior allogeneic transplantation and relapsed) and no active related infections (i.e., fungal or viral)
* In the case of allogeneic transplantation relapse, there should be no active acute graft-versus-host disease (GVHD) of any grade and no chronic GVHD other than mild skin, oral, or ocular GVHD not requiring systemic immunosuppression
* No known active brain metastases, other neurological disorders/dysfunction or history of seizure disorder, or other neurological dysfunction
* Karnofsky performance status 60-100%
* Life expectancy > 3 months
* Total bilirubin normal
* AST and ALT =< 2.5 times upper limit of normal
* Creatinine normal or creatinine clearance >= 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception during and for 3 months after the last dose of obatoclax mesylate
* At least 4 weeks since prior radiotherapy
* More than 2 days since prior steroids
* More than 2 weeks since prior low-dose chlorambucil
* WBC >= 3,000/mm^3
* ANC >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* At least 2 weeks since prior valproic acid

Exclusion Criteria:

* Uncontrolled concurrent medical condition or illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia including QTc > 450 msec
* Patients who are intolerant or refractory to prior treatment with bortezomib (refractory is defined as no response to prior treatment with bortezomib)
* Chemotherapy within the past 4 weeks (6 weeks for nitrosoureas or mitomycin C)
* Rituximab within the past 3 months (unless there is evidence of progression)
* Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Other concurrent investigational agents
* Combination antiretroviral therapy for HIV-positive patients
* No history of allergic reactions attributed to bortezomib, polyethylene glycol (PEG 300), or polysorbate 20
* No psychiatric illness or social situation that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-12; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of obatoclax mesylate when administered with bortezomib | 35 days
  Defined as the highest dose tested in which fewer than 33% of patients experienced DLT attributable to the study drug(s), when at least six patients were treated at that dose and are evaluable for toxicity. Graded according to the NCI CTCAE, Version 3.0.

SECONDARY OUTCOMES:
Toxicity as assessed by NCI CTCAE version 3.0 | Up to 26 weeks after completion of study treatment
  Summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity and nadir or maximum values for the laboratory measures, time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course.
Pharmacokinetics of obatoclax mesylate when administered with bortezomib | Dose 1 of course 1, pre-infusion, 1 and 2 hours into the infusion, immediately prior to the end of the infusion, then at 0.25, 0.5, 1, 2, 4, 8, 24, 48, 72, and 168 hours

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tuscano, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States